CLINICAL TRIAL: NCT06376409
Title: A Single-center, Prospective Study of Nutraceutical Supplements to Support Hair Growth in Females With Self-Perceived Thinning Hair
Brief Title: Prospective Study of Nutraceutical Supplements to Support Hair Growth in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceutical Wellness Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NW-HGN-02
Record Dates: First submitted 2024-04-11; First posted 2024-04-19 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Hair Thinning
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Single Group Assignment 6-month, single-center, prospective interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrafol Hair Growth Supplement (Experimental): 4 commercially available hair growth nutraceuticals will be evaluated. Treatment groups will be assigned according to the investigator's discretion. Efficacy comparisons will not be made across treatment groups.
  Interventions: Dietary Supplement: Nutrafol Women's Hair Growth Supplement; Dietary Supplement: Nutrafol Women's Balance Hair Growth Supplement; Dietary Supplement: Nutrafol Women's Vegan Hair Growth Supplement; Dietary Supplement: Nutrafol Women's Postpartum Hair Growth Supplement

INTERVENTIONS:
Dietary Supplement: Nutrafol Women's Hair Growth Supplement — Hair growth supplement for women ages 18 - 44
Dietary Supplement: Nutrafol Women's Balance Hair Growth Supplement — Hair growth supplement for women ages 45 - 70
Dietary Supplement: Nutrafol Women's Vegan Hair Growth Supplement — Hair growth supplement for women ages 18 - 44. This treatment group may also include subjects who do not follow a plant-based diet for purposes of extending the product claims beyond the initially studied demographic of women primarily adhering to a plant-based diet
Dietary Supplement: Nutrafol Women's Postpartum Hair Growth Supplement — Hair growth supplement for women ages 18 - 44. This product will be studied in the general women population and not postpartum women.

SUMMARY:
A single site open label interventional study evaluating currently marketed hair supplements targeting the underlying root causes of thinning hair.

DETAILED DESCRIPTION:
A single site open label interventional study evaluating currently marketed hair supplements targeting the underlying root causes of thinning hair. All treatment regimens are commercially available nutraceutical hair growth supplements. 45 subjects will be enrolled into each of the 4 supplement groups. Subjects will undergo a baseline, baseline + 48 hours, 90 day, 90 day + 48 hours, 180 day and 180 day + 48 hours visit and will have compliance phone calls at Days 45 and 135. All subject data will be compared to baseline in paired comparison for each subject using a historical control.

ELIGIBILITY:
Inclusion Criteria:

1. Females of all Fitzpatrick skin, and hair types between 18-70 years of age with self-perceived thinning, confirmed by a dermatologist.
2. Willing and able to adhere to the same dietary lifestyles for the duration of the study.
3. Able to understand and sign an informed consent agreement and photo release form approved by the Institutional Review Board
4. General good health, as determined by the Investigator or qualified sub-investigator.
5. Willing and able to attend all study visits and comply with the test product daily instructions.
6. Willing to use a mild non-medicated shampoo and conditioner for the duration of the study (medicated shampoo and conditioner refer to any prescription shampoo or conditioner as well as any over-the counter medicated shampoo or conditioner, such as those for treatment of dandruff or promoting hair growth).
7. Willing and able to cooperate with the requirements of the study.
8. Able to complete and understand the various questionnaires.

Exclusion Criteria:

1. Individuals who are pregnant, planning a pregnancy, nursing, or within 1-year post-partum.
2. Individuals who have experienced serious complications due to COVID-19 previously or during the study as determined by the investigator.
3. Clinical diagnosis of hair loss disorder such as alopecia areata, or scarring forms of alopecia.
4. Individuals who have had a history of any acute or chronic disease that could interfere with or increase the risk on study participation.
5. Individuals who have had a history of any acute or chronic medical or hair condition that could affect study results, such as a history of disordered eating.
6. Scalp hair loss on the treatment area, due to disease, injury, or medical therapy.
7. Current skin disease (e.g., psoriasis, atopic dermatitis, skin cancer, eczema, sun damage, seborrheic dermatitis), infection, cuts, and/ or abrasions on the scalp or condition (e.g., sunburn, tattoos) on the treatment area that, in the opinion of the Investigator or qualified sub-investigator, might put the subject at risk or interfere with the study conduct or evaluations.
8. History of surgical correction of hair loss on the scalp (i.e., hair transplant).
9. Use of any products or devices purported to promote scalp hair growth (e.g., finasteride or minoxidil) within the 6 months prior to the Baseline Visit.
10. Females who have recently (within the last 6 months) started the use of hormones for birth control or hormone replacement therapy (HRT). Women currently using hormones for birth control or HRT must have been on a stable dose (6 months or longer) in order to be eligible for the study (the initiation of HRT or birth control should not have been associated with the initiation of hair loss/thinning).
11. History of malignancy (except cutaneous squamous cell carcinoma and basal cell carcinoma) or currently undergoing chemotherapy or radiation treatments.
12. A known history of autoimmune thyroid disease, any other thyroid disorder/abnormality or other autoimmune disorders that in the opinion of the Investigator or qualified sub-investigator may interfere with the study treatment.
13. A known history of unstable or chronic depression or bipolar disease or any other condition that may impact the subject's participation in the opinion of the investigator or qualified sub-investigator.
14. A known allergy to any of the ingredients in the investigational product.
15. Utilization of low-level lasers for hair growth in the last three months.
16. Any condition that the Investigator thinks may put the subject at risk or interfere with their participation in the study or study results.
17. Known history of or current iron deficiency, bleeding disorders or platelet dysfunction syndrome as well as subjects receiving anticoagulant therapy or smokers with usage >20 cigarettes/day as reported by the subject.
18. Use of any medications or medicated shampoos that are known to potentially cause hair loss or affect hair growth, as determined by the Investigator or qualified sub-investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
The percent change in hair growth rate at Day 180 relative to baseline (Day 0) | 180 days
  The percent change in hair growth rate at Day 180 relative to baseline (Day 0) using Canfield HairMetrix® non-invasive device.

SECONDARY OUTCOMES:
The percent change in hair growth rate at Day 90 relative to baseline (Day 0) | 90 Days
  The percent change in hair growth rate at Day 90 relative to baseline (Day 0) as measured by the Canfield HairMetrix®.
The change in total hair count, terminal hairs, vellus hairs, anagen, and telogen hairs compared to baseline at 90 days | 90 days
  The change in total hair count, terminal hairs, vellus hairs, anagen, and telogen hairs compared to baseline at 90 days as measured by the Canfield HairMetrix® compared to baseline.
The change in total hair count, terminal hairs, vellus hairs, anagen, and telogen hairs compared to baseline at 180 days | 180 days
  The change in total hair count, terminal hairs, vellus hairs, anagen, and telogen hairs compared to baseline at 180 days as measured by the Canfield HairMetrix® compared to baseline.
The change in terminal to vellus ratio | 90 Days
  The change in terminal to vellus ratio as measured by the Canfield HairMetrix® at 90 days compared to baseline.
The change in terminal to vellus ratio | 180 Days
  The change in terminal to vellus ratio as measured by the Canfield HairMetrix® at 180 days compared to baseline.
The change in anagen to telogen ratio | 90 Days
  The change in terminal to vellus ratio per cm2 as measured by the Canfield HairMetrix® at 90 days compared to baseline.
The change in anagen to telogen ratio | 180 Days
  The change in terminal to vellus ratio per cm2 as measured by the Canfield HairMetrix® at 180 days compared to baseline.
The change in average number of hairs per follicular unit | 90 Days
  The change in average number of hairs per follicular unit as measured by the Canfield HairMetrix® at 90 days compared to baseline.
The change in average number of hairs per follicular unit | 180 Days
  The change in average number of hairs per follicular unit as measured by the Canfield HairMetrix® at 180 days compared to baseline.
The change in total hair width per cm2 | 90 Days
  The change in total hair width per cm2 as measured by the Canfield HairMetrix® at 90 days compared to baseline.
The change in total hair width per cm2 | 180 Days
  The change in total hair width per cm2 as measured by the Canfield HairMetrix® at 180 days compared to baseline.
The change in mean inter-follicular distance | 90 Days
  The change in mean inter-follicular distance as measured by the Canfield HairMetrix® at 90 days compared to baseline.
The change in mean inter-follicular distance | 180 Days
  The change in mean inter-follicular distance as measured by the Canfield HairMetrix® at 180 days compared to baseline.
Subjective assessments of change measured with Consumer Perception Questionnaire at 90 days | 90 Days
  Subjective assessments of change in hair growth and appearance measured with Consumer Perception Questionnaire at 90 days
Subjective assessments of change measured with Consumer Perception Questionnaire at 180 days | 180 Days
  Subjective assessments of change in hair growth and appearance measured with Consumer Perception Questionnaire at 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No